CLINICAL TRIAL: NCT06208579
Title: Feasibility and Effectiveness of Augmented Reality Assistance System for Pancreatic Surgery: a Prospective Study
Brief Title: Feasibility and Effectiveness of Augmented Reality Assistance System for Pancreatic Surgery
Acronym: ARAS-P
Status: Completed | Type: Observational
Sponsor: Klinikum Saarbrücken, Klinik für Allgemein-, Viszeral- und Thoraxchirurgie, Chirurgische Onkologie (Other)
Collaborators: Deutsches Forschungszentrum für Künstliche Intelligenz (DFKI) (Unknown); University of Kaiserslautern-Landau (Other)
Responsible Party: Principal Investigator, Dr.med Dr. habil Gregor A. Stavrou, Head of the Department, Klinikum Saarbrücken, Klinik für Allgemein-, Viszeral- und Thoraxchirurgie, Chirurgische Onkologie
Other Study IDs: 159/23
Record Dates: First submitted 2023-12-22; First posted 2024-01-17 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Pancreatectomy; Augmented Reality
Keywords: Augmented reality; Wearable devices; Pancreatic surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, resected pancreas specimen
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Pancreatic cancer necessitates surgical resection for complete tumor eradication, serving as the primary curative approach. However, pancreatic surgery is still challenging due to the organ's retroperitoneal anatomy and proximity to vital vascular systems. Thus, precise preparation and dissection of peripancreatic vessels are crucial during pancreatic surgery to reduce perioperative complications and improve oncological outcomes. The integration of preoperative computed tomography-derived reconstructed images, along with augmenting the resulting 3D model during surgical procedures, holds significant potential in this context. Augmented reality-assistance systems (ARAS) have seen use in various surgical fields, including orthopedic, plastic, and neurosurgery. Nevertheless, the application of ARAS in abdominal surgery has faced challenges related to organ shifting and deformities. The retroperitoneal nature of the pancreas, characterized by minimal intraoperative organ shifts and deformations, makes pancreatic surgery a promising candidate for ARAS. Despite this, there is a limited number of studies exploring the impact of ARAS during pancreatic surgery. Notably, existing investigations have primarily utilized augmented reality technology with 2D-display-based modalities. This prospective study aims to fill this gap by examining the usability, feasibility, and effectiveness of wearable ARAS during pancreatic surgery. By leveraging advanced technology seamlessly integrated into the surgical workflow, this research seeks to provide valuable insights into the practical application of ARAS, potentially enhancing the precision and outcomes of pancreatic surgery. The preliminary findings of this study will also be submitted for publication in a peer-reviewed journal.

ELIGIBILITY:
Inclusion Criteria:

* Patient consent
* Aged above 18 years
* Undergoing any type of pancreatectomy

Exclusion Criteria:

* Unresectable tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with any type of pancreatic tumor undergoing pancreatic surgery using an augmented reality-assistance system
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Rate of identified peripancreatic vessels with errors | During surgery

SECONDARY OUTCOMES:
User experience | Day 1
  User experience will be assessed using an adapted NASA Task Load Index (NASA-TLX, 5 questions, range, 1-10, with lower scores indicating lower cognitive workload)
Intraoperative blood loss | During surgery
Duration of operation | During surgery
Duration of hospital stay | Three months
Rate of tumor-free resection margin | One week
  Rate of tumor-free resection margin after pancreatic resection
Rate of morbidity | Three months
  Complications rate after pancreatic resection
Rate of mortality | Three months
  All cause death events

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Saarbrücken, Saarbrücken, Saarland, Germany

IPD SHARING:
Plan to Share IPD: No